CLINICAL TRIAL: NCT03310866
Title: Macintosh Laryngoscope Assisted Flexible Fiber Optic Endotracheal Intubation Versus Classic Fiber Optic Laryngoscope Alone Endotracheal Intubation for Modified Mallampati III&IV Patients : A Prospective Randomized Controlled Study
Brief Title: Macintosh Laryngoscope Assisted Fiberoptic Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R/17.08.102
Record Dates: First submitted 2017-10-05; First posted 2017-10-16 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Difficult Intubation
MeSH Terms: interventions — Optical Fibers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fiberoptic, airway (Active Comparator): Classical fiberoptic intubation assisted by side fenestrated airway and head tilt- chin lift- jaw thrust by 2 anesthetist
  Interventions: Device: fiberoptic, airway
- fiberoptic, Machintosh (Experimental): oral Fiberoptic bronchoscopic intubation assisted by Macintosh Laryngoscope, by 2 anesthetist
  Interventions: Device: fiberoptic, Machintosh

INTERVENTIONS:
Device: fiberoptic, airway — classic fiberoptic bronchoscope, fenstrated airway
  Arms: fiberoptic, airway
Device: fiberoptic, Machintosh — oral fiberoptic brochoscopic, Machintosh laryngoscope
  Arms: fiberoptic, Machintosh

SUMMARY:
During fiberoptic endotracheal intubation, the perfect airway exposure produced by the classic curved Macintosh laryngoscope in place of head tilt -chin lift-jaw thrust maneuver may increase the accuracy and produce rapid direct vocal cord access in a short time under Inhalation anesthesia to maintain the respiratory drive for grade III&VI Modified Mallampati .

DETAILED DESCRIPTION:
Managing difficult airway is critical for anesthesia-related morbidity and mortality. Fiberoptic laryngoscope is a reliable tool for endotracheal intubation in difficult airway cases (Modified Mallampatti III&IV), but always there is difficulty to visualize the glottis due to airway tendency to collapse, classically a specific fiberoptic airway with a side way is used and it may added head tilt chin lift jaw thrust. A new technique utilizing sevoflurane anesthesia to maintain the respiratory drive without exposing the patient to the stress of the awake airway instrumentation. Simultaneous utilization of both Macintosh curved laryngoscope and Fiberoptic bronchoscope during Endotracheal intubation (ETT) will be examined for the efficacy during difficult airway management.

All patients should be examined preoperatively for the scoring Modified Mallampati or non tongue protrusion mallampati (NT-MMT) airway score. The pharyngeal structures were then evaluated and the best view (lowest class) was recorded. The classification follows m-MMT and is as follows: class 1, full visibility of tonsils, uvula, and soft palate; class 2, visibility of hard and soft palate, upper portion of tonsils and uvula; class 3, visibility of the soft and hard palate and base of the uvula; and class 4, visibility of only the hard palate, class III or IV patients were included in the study. Inhalational anesthesia use maintains the respiratory drive of the patient allowing less stressful technique.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Modified Mallampati (NT-MMT) airway score III,VI
* American Society of Anaesthesiologists (ASA) physical class I-III
* Scheduled for elective cancer surgery under general anesthesia

Exclusion Criteria:

* Modified Mallampati I,II Airway scored patients.
* History of upper airway surgery.
* Patients with serious deformities of the mandible, maxilla, tongue, pharynx or larynx.
* Patients with a history of significant cardiac and pulmonary diseases,
* Obesity with BMI >40,
* Epilepsy, pregnancy, mental disease, neurological psychological disorders.
* Communication barrier.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
intubation time | during intubation
  time from introduction of the tip of the fiber optic laryngoscope till insertion of the tube in the laryngeal inlet down in the trachea in seconds.

SECONDARY OUTCOMES:
lower jaw relaxation | during intubation
  (Relaxed= 0, not fully=1, poor= 2)
Vocal cord position | during intubation
  (Abducted= 0, Intermediate opening= 1, Closed= 2)
Neck movements | during intubation and cuff inflation
  for endotracheal tube or cuff inflation (no=0, slight= 1, vigorous= 2),
Cough | during intubation and cuff inflation
  (absent= 0, present=1)
1st trial success rate | during intubation
  in percent
the number of trails | during intubation
  (1st trial=1, 2nd trial= 2, 3rd trial= 3)
mean arterial Blood pressure (MBP) | during intubation till 5 minutes after intubation
  basal, every minute during intubation, 1, 3, 5 minutes after intubation
mean heart rate (HR) | during intubation till 5 minutes after intubation
  basal, every minute during intubation, 1, 3, 5 minutes after intubation
desaturation (SpO2) | during intubation
  oxygen saturation <90% .(Yes=1, No= 0)

CONTACTS AND LOCATIONS:
Locations (1):
- Oncolgy Center, Mansoura University,, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
after publication
Supporting Information: SAP, CSR
Time Frame: no limit
Access Criteria: e mail mohamed.abdel_latif@yahoo.com